CLINICAL TRIAL: NCT02057835
Title: Safety, Tolerability and Pharmacokinetics of Single Rising Oral Doses of BI 691751 in Healthy Asian Male Volunteers in a Randomised, Double-blind, Placebo-controlled Design.
Brief Title: Safety, Tolerability and Pharmacokinetics of Single Rising Oral Doses of BI 691751 in Healthy Asian Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1334.5
Record Dates: First submitted 2014-02-06; First posted 2014-02-07 (Estimated); Results first posted 2015-12-16 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-11

CONDITIONS: Healthy

ARMS (4):
- BI 691751 low dose 1 (Experimental): BI 691751 low dose 1
  Interventions: Drug: Placebo to BI 691751; Drug: BI 691751 low dose 1
- BI 691751 low dose 2 (Experimental): BI 691751 low dose 2
  Interventions: Drug: Placebo to BI 691751; Drug: BI 691751 low dose 2
- BI 691751 middle dose (Experimental): BI 691751 middle dose
  Interventions: Drug: BI 691751 middle dose; Drug: Placebo to BI 691751
- BI 691751 high dose (Experimental): BI 691751 high dose
  Interventions: Drug: Placebo to BI 691751; Drug: BI 691751 high dose

INTERVENTIONS:
Drug: Placebo to BI 691751 — Placebo to BI 691751
  Arms: BI 691751 high dose
Drug: BI 691751 high dose — BI 691751 high dose
  Arms: BI 691751 high dose
Drug: BI 691751 middle dose — BI 691751 middle dose
  Arms: BI 691751 middle dose
Drug: Placebo to BI 691751 — Placebo to BI 691751
  Arms: BI 691751 low dose 1
Drug: BI 691751 low dose 1 — BI 691751 low dose 1
  Arms: BI 691751 low dose 1
Drug: Placebo to BI 691751 — Placebo to BI 691751
  Arms: BI 691751 low dose 2
Drug: Placebo to BI 691751 — Placebo to BI 691751
  Arms: BI 691751 middle dose
Drug: BI 691751 low dose 2 — BI 691751 low dose 2
  Arms: BI 691751 low dose 2

SUMMARY:
BI 691751 is currently being developed to inhibit growth and prevent rupture of atherosclerotic plaques and to consequently reduce the risk of major cardiovascular events in patients with established atherosclerotic disease. 1334.5 is a Pan Asian Phase 1 study to investigate safety, tolerability and pharmacokinetics of BI 691751 in healthy Chinese and Japanese male volunteers.

ELIGIBILITY:
Inclusion criteria:

1. Healthy males based upon a complete medical history, including a physical examination, vital signs (blood pressure, pulse rate), 12-lead ECG, and clinical laboratory tests
2. Chinese ethnicity, Japanese ethnicity according to the following criteria:

   Chinese; born in China or ethnic Chinese born outside of China, and a descendent of 4 ethnic Chinese grandparents who were all born in China Japanese; born in Japan and holding Japanese passport, have lived outside of Japan <10 years, and have parents and grandparents who were all born in Japan
3. Age within the range of 20 to 45 years
4. Body mass index within the range of 18.5 and 25 kg/m2
5. Signed and dated written informed consent prior to admission to the study in accordance with GCP and local legislation.

Exclusion criteria:

1. Any finding in the medical examination (including BP, PR or ECG) deviating from normal and judged clinically relevant by the investigator. Pulse rate outside the range of 50-90 bpm or blood pressure outside the ranges of 90-140 for systolic and 50-90 mmHg for diastolic blood pressure if confirmed by repeat measurement.
2. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
3. Any evidence of a concomitant disease judged clinically relevant by the investigator
4. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
5. Surgery of the gastrointestinal tract that could interfere with kinetics of the study drug
6. Diseases of the central nervous system (such as epilepsy), central neurological disorders or psychiatric disorders
7. History of relevant orthostatic hypotension, fainting spells, or blackouts
8. Relevant chronic or acute infections
9. History of relevant allergy/hypersensitivity (including allergy to the trial medication or its excipients)
10. Intake of drugs with a long half-life (greater than 24 hours) within 30 days or less than 10 half-lives of the respective drug prior to study drug administration
11. Use of drugs that might reasonably influence the results of the trial or that might prolong the QT/QTc interval within 14 days prior to study drug administration
12. Participation in another trial with investigational drug administration within 60 days prior to administration of trial medication
13. Smoker (more than 10 cigarettes or 3 cigars or 3 pipes/day)
14. Inability to refrain from smoking on specified trial days
15. Alcohol abuse (consumption of more than30 g/day)
16. Drug abuse or positive drug screen
17. Blood donation (more than 100 mL within 30 days prior to administration of trial medication or intended during the trial)
18. Intention to perform excessive physical activities within one week prior to administration of trial medication or during the trial
19. Inability to comply with dietary regimen of trial site
20. A marked baseline prolongation of QT/QTc interval (such as repeated demonstration of a QTc interval greater than 450 ms) or any other relevant ECG finding
21. A history of additional risk factors for Torsades de Pointes (such as heart failure, hypokalemia, or family history of Long QT Syndrome)
22. Subject is assessed by the investigator as unsuitable for inclusion, for instance, because considered not able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2014-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1334.5.82001 Boehringer Ingelheim Investigational Site, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Groups:
- Chinese: Placebo: Chinese participants received a single placebo tablet matching the BI 691751 tablets, orally with 240 mL water after an overnight fast of at least 10 hours.
- Chinese: BI 691751 5mg: Chinese participants received a single tablet of BI 691751 5mg orally with 240 mL water after an overnight fast of at least 10 hours.
- Chinese: BI 691751 10mg: Chinese participants received a single tablet of BI 691751 10mg orally with 240 mL water after an overnight fast of at least 10 hours.
- Chinese: BI 691751 30mg: Chinese participants received a single tablet of BI 691751 30mg orally with 240 mL water after an overnight fast of at least 10 hours.
- Chinese: BI 691751 60mg: Chinese participants received a single tablet of BI 691751 60mg orally with 240 mL water after an overnight fast of at least 10 hours.
- Japanese: Placebo: Japanese participants received a single placebo tablet matching the BI 691751 tablets, orally with 240 mL water after an overnight fast of at least 10 hours.
- Japanese: BI 691751 5mg: Japanese participants received a single tablet of BI 691751 5mg orally with 240 mL water after an overnight fast of at least 10 hours.
- Japanese: BI 691751 10mg: Japanese participants received a single tablet of BI 691751 10mg orally with 240 mL water after an overnight fast of at least 10 hours.
- Japanese: BI 691751 30mg: Japanese participants received a single tablet of BI 691751 30mg orally with 240 mL water after an overnight fast of at least 10 hours.
- Japanese: BI 691751 60mg: Japanese participants received a single tablet of BI 691751 60mg orally with 240 mL water after an overnight fast of at least 10 hours.
Period: Overall Study
Arm/Group | Chinese: Placebo | Chinese: BI 691751 5mg | Chinese: BI 691751 10mg | Chinese: BI 691751 30mg | Chinese: BI 691751 60mg | Japanese: Placebo | Japanese: BI 691751 5mg | Japanese: BI 691751 10mg | Japanese: BI 691751 30mg | Japanese: BI 691751 60mg
Started | 8 | 6 | 6 | 6 | 6 | 8 | 6 | 6 | 6 | 6
Completed | 8 | 4 | 6 | 6 | 6 | 8 | 6 | 6 | 6 | 6
Not Completed | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set which included all subjects who were documented to have taken study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Chinese: Placebo | Chinese: BI 691751 5mg | Chinese: BI 691751 10mg | Chinese: BI 691751 30mg | Chinese: BI 691751 60mg | Japanese: Placebo | Japanese: BI 691751 5mg | Japanese: BI 691751 10mg | Japanese: BI 691751 30mg | Japanese: BI 691751 60mg | Total
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6 | 8 | 6 | 6 | 6 | 6 | 64
Age, Continuous [Mean (Standard Deviation); unit: Years] | 25.3 (5.06) | 24.5 (3.73) | 23.0 (2.53) | 26.3 (4.55) | 28.8 (4.02) | 29.5 (3.82) | 31.7 (4.76) | 36.5 (2.74) | 31.0 (4.82) | 34.5 (0.84) | 29.0 (5.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 8 | 6 | 6 | 6 | 6 | 8 | 6 | 6 | 6 | 6 | 64

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Drug Related Adverse Events
Description: Percentage of participants with drug related adverse events (AEs)
Time Frame: From drug administration until 31 days after drug administration, 31 days
Population: Treated set
Measure: Number; unit: Percentage of participants
Arm/Group | Chinese: Placebo | Chinese: BI 691751 5mg | Chinese: BI 691751 10mg | Chinese: BI 691751 30mg | Chinese: BI 691751 60mg | Japanese: Placebo | Japanese: BI 691751 5mg | Japanese: BI 691751 10mg | Japanese: BI 691751 30mg | Japanese: BI 691751 60mg
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6 | 8 | 6 | 6 | 6 | 6
Percentage of participants | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

2. Secondary Outcome: Maximum Measured Concentration of the Analyte (Cmax)
Description: Maximum measured concentration of the analyte in plasma/whole blood
Time Frame: 1 hour (h) before drug administration and 20minutes (min), 40min, 1h, 1h 30min, 2h, 2h 30min, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 36h, 48h, 60h, 72h, 96h, 120h, 144h, 192h, 240h, 288h and 336h after drug administration
Population: All subjects of the treated set with the pharmacokinetic (PK) parameter calculated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Chinese: BI 691751 5mg | Chinese: BI 691751 10mg | Chinese: BI 691751 30mg | Chinese: BI 691751 60mg | Japanese: BI 691751 5mg | Japanese: BI 691751 10mg | Japanese: BI 691751 30mg | Japanese: BI 691751 60mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
nmol/L
  Plasma | 175 (45.7) | 477 (25.5) | 1450 (19.4) | 3690 (20.5) | 129 (33.2) | 421 (53.4) | 1520 (18.1) | 4270 (9.4)
  Blood | 247 (21.5) | 523 (19.7) | 1490 (22.1) | 3470 (16.4) | 213 (17.9) | 509 (35.4) | 1530 (22.4) | 3600 (12.4)

3. Secondary Outcome: Maximum Measured Concentration of the Analyte (Cmax) - Overall
Description: Maximum measured concentration of the analyte in plasma/whole blood for all participants (Chinese and Japanese)
Time Frame: as for outcome 2
Population: All subjects of the treated set with the pharmacokinetic (PK) parameter calculated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Groups:
- BI 691751 5mg: Participants received a single tablet of BI 691751 5mg orally with 240 mL water after an overnight fast of at least 10 hours.
- BI 691751 10mg: Participants received a single tablet of BI 691751 10mg orally with 240 mL water after an overnight fast of at least 10 hours.
- BI 691751 30mg: Participants received a single tablet of BI 691751 30mg orally with 240 mL water after an overnight fast of at least 10 hours.
- BI 691751 60mg: Participants received a single tablet of BI 691751 60mg orally with 240 mL water after an overnight fast of at least 10 hours.
Arm/Group | BI 691751 5mg | BI 691751 10mg | BI 691751 30mg | BI 691751 60mg
Number analyzed (Participants) | 12 | 12 | 12 | 12
nmol/L
  Plasma | 150 (41.4) | 448 (39.8) | 1490 (18.0) | 3970 (17.0)
  Blood | 229 (20.4) | 516 (27.2) | 1510 (21.2) | 3530 (14.0)

4. Secondary Outcome: Time From Dosing to the Maximum Measured Concentration of the Analyte (Tmax)
Description: Time from (last) dosing to the maximum measured concentration of the analyte in plasma/whole blood
Time Frame: as for outcome 2
Population: All subjects of the treated set with the pharmacokinetic (PK) parameter calculated.
Measure: Median (Full Range); unit: hours
Arm/Group | Chinese: BI 691751 5mg | Chinese: BI 691751 10mg | Chinese: BI 691751 30mg | Chinese: BI 691751 60mg | Japanese: BI 691751 5mg | Japanese: BI 691751 10mg | Japanese: BI 691751 30mg | Japanese: BI 691751 60mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
hours
  Plasma | 0.333 [0.333 to 0.667] | 0.667 [0.333 to 2.000] | 0.667 [0.333 to 1.000] | 0.667 [0.333 to 0.667] | 0.667 [0.333 to 0.667] | 0.500 [0.333 to 0.667] | 0.667 [0.333 to 0.667] | 0.667 [0.333 to 0.683]
  Blood | 0.333 [0.333 to 2.000] | 0.667 [0.333 to 2.000] | 0.667 [0.333 to 1.000] | 0.667 [0.333 to 0.667] | 0.500 [0.333 to 4.000] | 0.333 [0.333 to 0.667] | 0.667 [0.333 to 1.000] | 0.667 [0.333 to 0.683]

5. Secondary Outcome: Time From Dosing to the Maximum Measured Concentration of the Analyte (Tmax) - Overall
Description: Time from (last) dosing to the maximum measured concentration of the analyte in plasma/whole blood for all participants (Chinese and Japanese)
Time Frame: as for outcome 2
Population: All subjects of the treated set with the pharmacokinetic (PK) parameter calculated.
Measure: Median (Full Range); unit: hours
Arm/Group | BI 691751 5mg | BI 691751 10mg | BI 691751 30mg | BI 691751 60mg
Number analyzed (Participants) | 12 | 12 | 12 | 12
hours
  Plasma | 0.500 (41.4) [0.333 to 0.667] | 0.667 (39.8) [0.333 to 2.000] | 0.667 (18.0) [0.333 to 1.000] | 0.667 (17.0) [0.333 to 0.683]
  Blood | 0.333 (20.4) [0.333 to 4.000] | 0.500 (27.2) [0.333 to 2.000] | 0.667 (21.2) [0.333 to 1.000] | 0.667 (14.0) [0.333 to 0.683]

6. Secondary Outcome: Area Under the Concentration-time Curve of the Analyte Over the Time Interval From 0 Extrapolated to Infinity (AUC0-infinity)
Description: Area under the concentration-time curve of the analyte in plasma/whole blood over the time interval from 0 extrapolated to infinity (AUC0-infinity)
Time Frame: as for outcome 2
Population: All subjects of the treated set with the pharmacokinetic (PK) parameter calculated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | Chinese: BI 691751 5mg | Chinese: BI 691751 10mg | Chinese: BI 691751 30mg | Chinese: BI 691751 60mg | Japanese: BI 691751 5mg | Japanese: BI 691751 10mg | Japanese: BI 691751 30mg | Japanese: BI 691751 60mg
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 6
nmol*h/L
  Plasma (N=0,5,6,6,0,0,6,6) | NA (NA) — gMean and gCV were not calculated as the concentrations were not quantifiable at the terminal phase and this parameter could not be evaluated in most of subjects. | 5280 (17.3) | 18000 (22.3) | 37400 (23.9) | NA (NA) — gMean and gCV were not calculated as the concentrations were not quantifiable at the terminal phase and this parameter could not be evaluated in most of subjects. | NA (NA) — gMean and gCV were not calculated, since, according to internal rules, descriptive statistics were considered as reliable only when data from at least 2/3 of the subjects were available. | 22400 (28.0) | 42000 (14.1)
  Blood (N=5,6,6,6,6,6,6,6) | 31600 (23.3) | 51800 (22.4) | 75600 (13.5) | 118000 (10.3) | 35600 (65.5) | 48700 (19.6) | 91800 (38.6) | 105000 (11.4)

7. Secondary Outcome: Area Under the Concentration-time Curve of the Analyte Over the Time Interval From 0 Extrapolated to Infinity (AUC0-infinity) - Overall
Description: Area under the concentration-time curve of the analyte in plasma/whole blood over the time interval from 0 extrapolated to infinity for all participants (Chinese and Japanese)
Time Frame: as for outcome 2
Population: All subjects of the treated set with the pharmacokinetic (PK) parameter calculated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | BI 691751 5mg | BI 691751 10mg | BI 691751 30mg | BI 691751 60mg
Number analyzed (Participants) | 11 | 12 | 12 | 12
nmol*h/L
  Plasma (N=0, 8, 12, 12) | NA (NA) — gMean and gCV were not calculated as the concentrations were not quantifiable at the terminal phase and this parameter could not be evaluated in most of subjects. | 5210 (27.8) | 20100 (26.8) | 39600 (19.6)
  Blood (N=11, 12, 12, 12) | 33800 (47.5) | 50200 (20.4) | 83300 (29.2) | 112000 (12.1)

8. Secondary Outcome: Area Under the Concentration-time Curve of the Analyte Over the Time Interval From 0 to the Time of the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of the analyte in plasma/whole blood over the time interval from 0 to the time of the last quantifiable data point (AUC0-tz)
Time Frame: as for outcome 2
Population: All subjects of the treated set with the pharmacokinetic (PK) parameter calculated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | Chinese: BI 691751 5mg | Chinese: BI 691751 10mg | Chinese: BI 691751 30mg | Chinese: BI 691751 60mg | Japanese: BI 691751 5mg | Japanese: BI 691751 10mg | Japanese: BI 691751 30mg | Japanese: BI 691751 60mg
Number analyzed (Participants) | 4 | 6 | 6 | 6 | 6 | 6 | 6 | 6
nmol*h/L
  Plasma | 1320 (22.1) | 4720 (17.8) | 17500 (23.1) | 37000 (24.2) | 1310 (27.3) | 5060 (38.7) | 21600 (28.6) | 41100 (13.8)
  Blood | 19200 (11.9) | 27900 (9.9) | 41000 (14.6) | 66600 (14.2) | 19500 (22.2) | 29600 (11.1) | 48300 (16.2) | 66800 (9.5)

9. Secondary Outcome: Area Under the Concentration-time Curve of the Analyte Over the Time Interval From 0 to the Time of the Last Quantifiable Data Point (AUC0-tz) - Overall
Description: Area under the concentration-time curve of the analyte in plasma/whole blood over the time interval from 0 to the time of the last quantifiable data point (AUC0-tz) for all participants (Chinese and Japanese)
Time Frame: as for outcome 2
Population: All subjects of the treated set with the pharmacokinetic (PK) parameter calculated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | BI 691751 5mg | BI 691751 10mg | BI 691751 30mg | BI 691751 60mg
Number analyzed (Participants) | 10 | 12 | 12 | 12
nmol*h/L
  Plasma (N=10, 12, 12, 12) | 1310 (23.9) | 4890 (28.7) | 19500 (27.2) | 39000 (19.6)
  Blood (N=10, 12, 12, 12) | 19400 (17.9) | 28700 (10.5) | 44500 (17.1) | 66700 (11.5)

10. Secondary Outcome: Terminal Half-life of the Analyte (T1/2)
Description: Terminal half-life (T1/2) of the analyte in plasma/whole blood
Time Frame: as for outcome 2
Population: All subjects of the treated set with the pharmacokinetic (PK) parameter calculated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Chinese: BI 691751 5mg | Chinese: BI 691751 10mg | Chinese: BI 691751 30mg | Chinese: BI 691751 60mg | Japanese: BI 691751 5mg | Japanese: BI 691751 10mg | Japanese: BI 691751 30mg | Japanese: BI 691751 60mg
Number analyzed (Participants) | 5 | 5 | 6 | 6 | 6 | 6 | 6 | 6
hours
  Plasma (N=0,5,6,6,0,0,6,6) | NA (NA) — gMean and gCV were not calculated as the concentrations were not quantifiable at the terminal phase and this parameter could not be evaluated in most of subjects. | 94.6 (29.8) | 102 (34.3) | 73.5 (40.4) | NA (NA) — gMean and gCV were not calculated as the concentrations were not quantifiable at the terminal phase and this parameter could not be evaluated in most of subjects. | NA (NA) — gMean and gCV were not calculated as the concentrations were not quantifiable at the terminal phase and this parameter could not be evaluated in most of subjects. | 95.0 (64.7) | 89.9 (26.2)
  Blood (N=5,6,6,6,6,6,6,6) | 243 (40.6) | 333 (30.6) | 393 (23.1) | 417 (23.7) | 290 (62.8) | 265 (26.2) | 403 (48.9) | 340 (26.0)

11. Secondary Outcome: Terminal Half-life of the Analyte (T1/2) - Overall
Description: Terminal half-life (T1/2) of the analyte in plasma/whole blood for all participants (Chinese and Japanese)
Time Frame: as for outcome 2
Population: All subjects of the treated set with the pharmacokinetic (PK) parameter calculated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | BI 691751 5mg | BI 691751 10mg | BI 691751 30mg | BI 691751 60mg
Number analyzed (Participants) | 11 | 12 | 12 | 12
hours
  Plasma (N=0, 8, 12, 12) | NA (NA) — gMean and gCV were not calculated as the concentrations were not quantifiable at the terminal phase and this parameter could not be evaluated in most of subjects. | 84.2 (28.9) | 98.4 (48.4) | 81.3 (34.1)
  Blood (N=11, 12, 12, 12) | 267 (51.6) | 297 (29.8) | 398 (35.9) | 377 (26.2)

ADVERSE EVENTS:
Time Frame: From drug administration until 31 days after drug administration, 31 days
Groups:
- Placebo: Participants received a single placebo tablet matching the BI 691751 tablets, orally with 240 mL water after an overnight fast of at least 10 hours.
Arm/Group | Placebo | BI 691751 5mg | BI 691751 10mg | BI 691751 30mg | BI 691751 60mg
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/12 | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 6/16 | 6/12 | 4/12 | 3/12 | 7/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=16) | BI 691751 5mg (N=12) | BI 691751 10mg (N=12) | BI 691751 30mg (N=12) | BI 691751 60mg (N=12)
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 1 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1
Liver function test abnormal (Investigations) | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 2 | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 2 | 3 | 2
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 2
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0 | 2
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.